CLINICAL TRIAL: NCT04176224
Title: Clinical Pharmacology Study of Oral Edaravone in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Clinical Pharmacology Study of Oral Edaravone in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MT-1186-J04
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Japanese Patients With ALS
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MT-1186 (Experimental): Patients receive the edaravone oral suspension.
  Interventions: Drug: MT-1186

INTERVENTIONS:
Drug: MT-1186 — Suspension
  Other Names: Edaravone

SUMMARY:
To evaluate the pharmacokinetics of single doses of edaravone oral suspension in Patients with Amyotrophic Lateral Sclerosis

ELIGIBILITY:
Inclusion Criteria:

The key criteria are listed below.

* Patients aged between 20 and 75 years at the time of informed consent
* Japanese patients
* Among patients with ALS, those "Clinically definite ALS," "Clinically probable ALS" or "Clinically probable-laboratory-supported ALS" according to El Escorial Revised Airlie House criteria
* Patients who can consent to contraception
* Patients who have thoroughly understood the contents of the study and voluntarily provided written informed consent to participate in the study

Exclusion Criteria:

The key criteria are listed below.

* Patients in whom the possibility could not be ruled out that the current symptoms were symptoms of a disease requiring differential diagnosis, such as cervical spondylosis and multifocal motor neuropathy
* Patients undergoing treatment for malignancy
* Patients who have presence of clinically significant liver, heart, or renal disease requiring hospitalization (except ALS) and infections requiring antibiotics. Patients who have a problem in general condition and are judged ineligible by the Investigator
* Body mass index (BMI) of <18.0 or >30.0, or a body weight of <50 kg
* Patients judged by the investigator (or subinvestigator) to be unsuitable for the study for any other reason

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shimizu H, Nishimura Y, Shiide Y, Akimoto M, Yashiro M, Ueda M, Hirai M, Yoshino H, Mizutani T, Kanai K, Kano O, Kimura H, Sekino H, Ito K. Pharmacokinetics of Edaravone Oral Suspension in Patients With Amyotrophic Lateral Sclerosis. Clin Ther. 2023 Dec;45(12):1251-1258. doi: 10.1016/j.clinthera.2023.09.025. Epub 2023 Nov 11. PMID 37953075

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-1186: ALS patients receive the edaravone oral suspension.
Period: Overall Study
Arm/Group | MT-1186
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MT-1186
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero up to the Last Quantifiable Concentration Time-point (AUC0-t) of Unchanged Edaravone
Time Frame: Plasma samples are collected: Day 1 at pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, and 12 hours; Day 2 at 24 hours after administration.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | MT-1186
Number analyzed (Participants) | 9
ng·h/mL | 1719 (808)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MT-1186
Number analyzed (Participants) | 9
ng/mL | 1903 (978.5)

3. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | MT-1186
Number analyzed (Participants) | 9
h | 0.25 [0.08 to 0.50]

4. Primary Outcome: Terminal Elimination Half-life (t1/2) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | MT-1186
Number analyzed (Participants) | 9
h | 6.11 (1.17)

5. Primary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | MT-1186
Number analyzed (Participants) | 9
1/h | 0.118 (0.028)

6. Primary Outcome: Mean Residence Time (MRT) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | MT-1186
Number analyzed (Participants) | 9
h | 2.14 (0.52)

7. Primary Outcome: Apparent Total Clearance (CL/F) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MT-1186
Number analyzed (Participants) | 9
L/h | 72.5 (33.4)

8. Primary Outcome: Apparent Distribution Volume at Elimination Phase (Vz/F) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MT-1186
Number analyzed (Participants) | 9
L | 603 (196)

9. Primary Outcome: Apparent Distribution Volume at Steady State (Vss/F) of Unchanged Edaravone
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MT-1186
Number analyzed (Participants) | 9
L | 155.7 (85.0)

10. Primary Outcome: Cumulative Amount of Drug Excreted in Urine From Time Zero up to 24 Hours (Ae0-24) of Unchanged Edaravone
Time Frame: Urine samples are collected: 0 to 24 hours after oral administration
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MT-1186
Number analyzed (Participants) | 9
mg | 0.534 (0.110)

11. Primary Outcome: Cumulative Percentage of Drug Excreted in Urine From Time Zero up to 24 Hours (Ae0-24) of Unchanged Edaravone
Time Frame: Urine samples are collected: 0 to 24 hours after oral administration
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MT-1186
Number analyzed (Participants) | 9
percentage | 0.508 (0.105)

12. Primary Outcome: Renal Clearance (CLr) of Unchanged Edaravone
Time Frame: Urine samples are collected: 0 to 24 hours after oral administration
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MT-1186
Number analyzed (Participants) | 9
L/h | 0.374 (0.232)

13. Secondary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: Day 1 to 8
Measure: Count of Participants; unit: Participants
Arm/Group | MT-1186
Number analyzed (Participants) | 9
Participants
  Number of Participants with Adverse events | 1
  Number of Participants with adverse drug reactions | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 8
Arm/Group | MT-1186
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-1186 (N=9)
Blood urine present (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04176224/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT04176224/SAP_001.pdf